CLINICAL TRIAL: NCT01462136
Title: A Phase 1 Study To Assess The Pharmacokinetics, Safety, And Tolerability of Intravenous ACHN-490 Injection in Volunteers With Varying Degrees of Renal Dysfunction Compared to Healthy Volunteers
Brief Title: PK Study of ACHN-490 Injection in Renally Impaired Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achaogen, Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACHN-490-004
Record Dates: First submitted 2011-09-09; First posted 2011-10-31 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Renal Insufficiency
Keywords: PK study
MeSH Terms: conditions — Renal Insufficiency | interventions — plazomicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACHN-490 Injection (Experimental)
  Interventions: Drug: ACHN-490 Injection

INTERVENTIONS:
Drug: ACHN-490 Injection — 7.5 mg/kg single dose administered intravenously over 30 minutes

SUMMARY:
The purposes of this study is to assess the relationship between renal function and pharmacokinetics of ACHN-490 Injection.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between 18 and 75 years of age and with a body mass index ≥ 19 to ≤ 32 kg/m2, and weight of ≥ 40 kg.
2. Normal renal function (Group I), or pre-existing renal impairment (Groups II- IV). The disease process responsible for the underlying renal dysfunction must be stable at the time of study entry, and the subject cannot have had episodes of acute renal disease in the year prior to dosing.
3. Two CrCl determinations obtained during the screening portion of the study, with the lower value within 25% of the higher value.
4. Females of child-bearing potential (defined as less than one year post-menopause) are eligible for enrollment if they are not breast feeding, they have a negative serum pregnancy test before study entry, and they are willing to use a highly effective method of contraception* for at least three months before study drug administration, during the study, and for at least one month after study completion.
5. Subjects in stable health as judged by the investigator based on the laboratory criteria and no clinically significant findings on the medical history or physical examination.
6. Subjects who are willing to comply with all study activities and procedures and have provided written informed consent prior to any study procedures and have signed and dated a HIPAA authorization form.

Exclusion Criteria:

1. Subjects requiring hemodialysis or peritoneal dialysis
2. Unstable cardiovascular disease,
3. Uncontrolled hypertension, asthma, diabetes (type I or type II), thyroid disease, or seizure disorder.
4. Myasthenia gravis, or any other neuromuscular disorder.
5. Known infection with Hepatitis B (antigen positive), Hepatitis C (antibody positive), or HIV.
6. Active malignancy; carcinoma in situ of the prostate or the skin (basal cell or squamous cell) are permitted.
7. Presence of functioning transplant organ or blood procedure.
8. Significant change in either over-the-counter or prescription medications or supplements within the two weeks prior to dosing, defined as any new medication or any dosage adjustment that is significant in the judgment of the investigator and the medical monitor.
9. Use of drugs known to cause renal disease such as non-steroidal anti-inflammatory drugs in the two weeks prior to dosing.
10. History of significant hearing loss or a family history of hearing loss, excluding age related (≥ age 65) hearing loss. A prior diagnosis of sensorineural hearing loss or Ménière's disease.
11. Clinically significant illness, including viral syndromes within three weeks of dosing.
12. Current participation in a clinical study of an investigational product.
13. Taken any investigational medication/therapy within 30 days or 5 half-lives, whichever is longer, before dosing of ACHN-490 Injection.
14. Consumed more than 28 units of ethanol per week at any time in the 6 months before dosing (1 unit of ethanol is equivalent to 8 ounces of beer, 4 ounces of wine, or 1 ounce of spirits) or history of alcoholism and/or drug/chemical abuse. Also, consumption of any amount of ethanol within 48 hours of ACHN-490 Injection dosing.
15. Donated more than 500 mL of blood within 60 days prior to signing the informed consent form.
16. Previous participation in this or any other ACHN-490 Injection study.
17. Known hypersensitivity to Aminoglycosides or any component of the ACHN-490 Injection.
18. Any other medical, psychological, or social condition which, in the opinion of the principal investigator (PI) or the medical monitor, would prevent the subject from fully participating in the study, would represent a concern for study compliance or would constitute a safety concern to the subject.
19. An employee of the investigator or study center with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, or a family member of the employee or investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09

PRIMARY OUTCOMES:
Composite of Pharmacokinetics | 0-96 hours
  Plasma PK parameters, including area under the curve from time zero to the last quantifiable sample (AUC0-t) and also extrapolated to infinity (AUC0-∞) total clearance (CLT), steady-state volume of distribution (Vss), maximum concentration (Cmax), time to maximum plasma concentration (Tmax), and the terminal-phase half life (t1/2)
  Urine PK including renal clearance (CLR), fraction of drug excreted in the urine expressed as a percentage of the ACHN-490 dose administered (Ae%), and amount of drug excreted in the urine through 24 hours (Ae0-24) and through 48 hours (Ae0-48).

SECONDARY OUTCOMES:
Safety | Days 1 to 14
  Safety and tolerability, including adverse events (AEs), and incidence and magnitude of clinically significant changes from baseline in clinical laboratory values (hematology, chemistry, and urinalysis), physical examination, and electrocardiogram (ECG).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Achaogen, Inc.

REFERENCES:
- [Derived] Komirenko AS, Riddle V, Gibbons JA, Van Wart S, Seroogy JD. A Phase 1 Study To Assess the Pharmacokinetics of Intravenous Plazomicin in Adult Subjects with Varying Degrees of Renal Function. Antimicrob Agents Chemother. 2018 Nov 26;62(12):e01128-18. doi: 10.1128/AAC.01128-18. Print 2018 Dec. PMID 30275092